CLINICAL TRIAL: NCT03065153
Title: Interaction Between Trunk and Gait Performance in Both Healthy Adults and Stroke Patients
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Rehabilitation Hospital RevArte (Unknown)
Responsible Party: Principal Investigator, Tamaya Van Criekinge, Principal Investigator, Universiteit Antwerpen
Other Study IDs: TVC-2
Record Dates: First submitted 2017-02-13; First posted 2017-02-27 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Healthy; Gait, Hemiplegic
Keywords: Torso; Trunk
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy individuals without any neurological or orthopaedic disorder that could influence motor performance and balance
- Stroke: Individuals suffered from a haemorrhagic or ischaemic stroke. Diagnosis has to be confirmed on the basis of CT or MRI imaging.

SUMMARY:
The aim is to investigate the biomechanical interaction between trunk and gait performance in both healthy and stroke subjects. People after stroke often have an impaired trunk function, resulting in balance and gait disorders. Pathological movement patterns after stroke can be compared with normative data as motion capture systems provide more sensitive data to explore the interaction between trunk performance and gait in contrast to the clinical measures used in literature.

DETAILED DESCRIPTION:
Evidence has shown that trunk performance is related to measures of balance, gait and functional ability. Yet, several aspects of trunk performance such as sitting balance, trunk muscle strength, selective trunk movements and trunk position sense are impaired after stroke. This implies that impaired trunk performance will inevitably lead to impaired postural control during activities performed while standing and walking. Nonetheless, the interaction between increased trunk performance and improvements in activities performed while standing and walking is not evident. It has previously been stated that therapy primarily induces treatment effects on the abilities at which training is specifically aimed. However, previous research has shown that additional trunk exercises improve not only trunk performance but also standing balance and mobility. Yet, the clinical outcome measures used in previous studies are not suitable to explore the relationship between trunk and gait performance and cannot explain the underlying mechanisms of the therapeutic effects. Since studies using sensitive motion analyses to investigate trunk biomechanics during gait are sparse in both healthy subjects and subjects with stroke. Data will be gathered by a Vicon analysis system (©Vicon Motion Systems Ltd., London, UK) with a measuring frequency of 100 Hz and eight infrared automated cameras (Vicon T10 cameras, 100 fps, 1 Megapixel) measured the 3D coordinates of the reflective markers. In addition, initial contact and toe off were defined based on the ankle trajectories of the reflective markers together with 3 AMTI type OR 6-7 force plates (1000 fps, 46x50x8 cm) and 1 AccuGait® (1000 fps) force plate recordings. Reflective motion trackers were attached to anatomical landmarks on the participant's body according to the standard Plug-In-Gait model. Furthermore, a 16 channel telemetric wireless EMG system (Arion Zerowire) will measure muscle activity.

ELIGIBILITY:
Inclusion Criteria Stroke:

1. haemorrhagic or ischaemic stroke diagnosis, confirmed on the basis of CT or MRI imaging;
2. no known history of previous stroke;
3. stroke onset within five months;
4. patients are between 18 and 85 years of age;

Exclusion Criteria Stroke:

1. A score of 20 or higher on the Trunk Impairment Scale which indicates normal truncal function;
2. A score lower than two on the Functional Ambulation Categories (FAC) as patients needed to be able to ambulate without physical support to ensure that gait analysis can be executed safely;
3. Not able to sit independently for 30 seconds on a stable surface;
4. They suffer from other neurological and orthopaedic disorders that could influence motor performance and balance;
5. not able to understand instructions.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers: community sample Stroke: Rehabilitation Hospital RevArte, primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Continous relative phase (of the trunk) by means of 3D full body gait analysis | Once, in the week of inclusion
  Phase difference of the upper and lower trunk in the transverse plane which assesses trunk coordination

SECONDARY OUTCOMES:
Lateral trunk displacements by means of 3D full body gait analysis (mm) | Once, in the week of inclusion
  Medio-lateral movements of the upper and lower trunk in the frontal plane
Vertical trunk displacements by means of 3D full body gait analysis (mm) | Once, in the week of inclusion
  Up- and downward movements of the upper and lower trunk in the frontal plane
Anteroposterior trunk displacements by means of 3D full body gait analysis (mm) | Once, in the week of inclusion
  Forward and backward movements of the upper and lower trunk in the sagittal plane

OTHER OUTCOMES:
Walking speed | Once, in the week of inclusion
  (m/s)
Step length | Once, in the week of inclusion
  (m)
Step time | Once, in the week of inclusion
  (s)
Step width | Once, in the week of inclusion
  (m)
% stance | Once, in the week of inclusion
Erector Spinae muscle activity (EMG) | Once, in the week of inclusion
  The amplitude and timing of muscle contractions

CONTACTS AND LOCATIONS:
Overall Officials: Steven Truijen, Prof. Dr., Study Chair — Universiteit Antwerpen
Locations (1):
- RevArte Rehabilitation Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided